CLINICAL TRIAL: NCT07081009
Title: Evaluation of the Incidence and Risk Factors of Myocardial Injury After Noncardiac Surgery (MINS) in Lumbar Surgery Patients
Brief Title: Myocardial Injury After Noncardiac Surgery (MINS) in Lumbar Surgery Patients
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Mehmet sahap, asist prof, Ankara City Hospital Bilkent
Other Study IDs: mıns and lumbar surgery
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-07

CONDITIONS: MYOCARD INFARCTUS; Non Cardiac Surgery; Lumbar Surgery; Anesthesia
Keywords: Myocardial injury; noncardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 270 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mins positivity: Patients with high sensitive troponin positivity after surgery
- Mins Negative: Patients with negative high sensitive troponin after surgery

SUMMARY:
The aim of this study is to evaluate the incidence of myocardial injury after noncardiac surgery (MINS) in patients undergoing lumbar surgery, and to investigate the associated risk factors.

ELIGIBILITY:
Inclusion criteria Age ≥18 years Elective lumbar stabilization surgery

Exclusion criteria History of cardiac surgery Recent acute MI (<30 days) Chronic elevated troponin levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 180 patients aged 18 years and older who are scheduled to undergo elective lumbar stabilization will be included. Participants will be enrolled upon physician approval and informed consent.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
1. Ischemia-related myocardial damage after noncardiac surgery | After surgery 30 days
  Ischemia-related myocardial damage occurring within 30 days after noncardiac surgery

SECONDARY OUTCOMES:
2. Causes of myocardial damage due to ischemia following noncardiac surgery | 30 days
  To identify risk factors for myocardial damage due to ischemia following noncardiac surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to the inadequate database network, patient information will not be shared with third parties. Patient data may be shared with journals upon request.